CLINICAL TRIAL: NCT02371941
Title: A Randomized, Double-blind, Placebo-controlled Study of the Use of Oral Cromolyn Sodium for the Treatment of Eosinophilic Esophagitis
Brief Title: Oral Cromolyn Sodium for the Treatment of Eosinophilic Esophagitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Tennessee (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 13-02521-FB
Record Dates: First submitted 2015-02-11; First posted 2015-02-26 (Estimated); Results first posted 2023-10-26 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: Eosinophilic Esophagitis
MeSH Terms: conditions — Eosinophilic Esophagitis | interventions — Cromolyn Sodium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oral cromolyn (Experimental): Subjects randomized to the experimental arm will receive oral cromolyn sodium. The dose will be per current package insert for oral cromolyn:
  Subjects 2-12 years of age - 100 mg (1 ampule) 4 times daily Subjects 13-18 years of age - 200 mg (2 ampules) 4 times daily
  Interventions: Drug: oral cromolyn sodium
- Placebo (Placebo Comparator): Subjects randomized to placebo will receive normal saline ampules Subjects 2-12 years of age - 1 ampule 4 times daily Subjects 13-18 years of age - 2 ampules 4 times daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: oral cromolyn sodium — Oral cromolyn sodium
  Other Names: Gastrocrom
  Arms: Oral cromolyn
Drug: Placebo — Saline
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled study of oral cromolyn sodium when made into a viscous preparation for the treatment of eosinophilic esophagitis.

DETAILED DESCRIPTION:
Eosinophilic esophagitis is an antigen-mediated allergic disease of the esophagus characterized by symptoms of gastrointestinal complaints and eosinophilic inflammation limited to the esophagus. Currently, first line therapeutic recommendations include swallowed, topical steroids or dietary therapy. While both work for the majority of patients, they both have limitations.

The investigators are examining the use of oral cromolyn sodium as a treatment for this condition. This medication is a non-steroid that is already approved for other conditions. When taken orally, it is essentially not absorbed systemically, so side effects are minimal. There is only 1 brief, retrospective report of its use in this condition suggesting it does not work. However, from studying swallowed, topical steroids, it may require formulating the medication into a viscous preparation for it to work.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of eosinophilic esophagitis

Exclusion Criteria:

* Concomitant treatment with swallowed corticosteroids. Any prior use of swallowed corticosteroids will require a 4 week washout period.
* Pregnancy (all females of child bearing potential will have urine pregnancy test done at baseline).
* Evidence of pathologic eosinophilia in other locations in the GI tract.
* Participation in another research protocol
* Reduced Renal or Hepatic Function (all subjects will have a baseline creatinine and liver function panel drawn)

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 16 (Actual)
Dates: Start 2014-12; Primary Completion 2017-07 (Actual); Study Completion 2017-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jay A Lieberman, MD, Principal Investigator — The University of Tennessee Health Science Center
Locations (1):
- LeBonheur Children's Hospital, Memphis, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lieberman JA, Zhang J, Whitworth J, Cavender C. A randomized, double-blinded, placebo-controlled study of the use of viscous oral cromolyn sodium for the treatment of eosinophilic esophagitis. Ann Allergy Asthma Immunol. 2018 May;120(5):527-531. doi: 10.1016/j.anai.2018.03.006. Epub 2018 Mar 12. PMID 29544738

RESULTS

PARTICIPANT FLOW:
Groups:
- Oral Cromolyn: Subjects randomized to the experimental arm will receive oral cromolyn sodium. The dose will be per current package insert for oral cromolyn:
  Subjects 2-12 years of age - 100 mg (1 ampule) 4 times daily Subjects 13-18 years of age - 200 mg (2 ampules) 4 times daily
  oral cromolyn sodium: Oral cromolyn sodium
Period: Overall Study
Arm/Group | Oral Cromolyn | Placebo
Started | 9 | 7
Completed | 9 | 6
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Oral Cromolyn | Placebo | Total
Number analyzed (Participants) | 9 | 7 | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 9 | 7 | 16
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.4 (4.1) | 12.8 (4) | 11.5 (4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 3 | 8
  Male | 4 | 4 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 8 | 7 | 15
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 9 | 7 | 16

OUTCOME MEASURES:

1. Primary Outcome: Peak Esophageal Eosinophil Count
Description: Measure of the peak esophageal eosinophil count on esophageal biopsy specimens after 2 months of therapy
Time Frame: 2 months
Measure: Median (Standard Deviation); unit: Peak # of eosinophils counted per field
Arm/Group | Oral Cromolyn | Placebo
Number analyzed (Participants) | 9 | 6
Peak # of eosinophils counted per field | 57.3 (44.02) | 71.3 (52.7)

2. Secondary Outcome: Symptoms as Measured by Pediatric Eosinophilic Esophagitis Symptom Score
Description: Symptom scores will be measures at baseline, 1 month, and 2 months using a symptom scoring assessment tool known as the Pediatric Eosinophilic Esophagitis Symptom Score (PEESS).
  The PEESS is a validated symptom score that is completed by the parent of the patient.
  It encompasses frequency and severity of EoE related symptoms over the past month.
  The minimum score = 0. The max score = 98 The higher the score/value, the more severe and/or frequent the symptoms and therefore a worse outcome.
Time Frame: Baseline as compared to 2 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Oral Cromolyn | Placebo
Number analyzed (Participants) | 9 | 6
units on a scale
  Baseline PEES score | 37.89 (12.2) | 30.3 (13.7)
  2 month PEES score | 17.5 (12.8) | 22.3 (19.1)

ADVERSE EVENTS:
Time Frame: 2 months
Arm/Group | Oral Cromolyn | Placebo
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/7
Other Adverse Events (participants affected / at risk) | 8/9 | 4/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oral Cromolyn (N=9) | Placebo (N=7)
nausea (Gastrointestinal disorders) | 5 (5) | 1 (1)
abdominal pain (Gastrointestinal disorders) | 4 (4) | 2 (2)
headache (Nervous system disorders) | 4 (4) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-03-10): https://cdn.clinicaltrials.gov/large-docs/41/NCT02371941/Prot_SAP_000.pdf